CLINICAL TRIAL: NCT02016638
Title: Sleep Quality in Pregnancy and Its Impact on Pregnancy Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, S.K.SHARMA, Professor and Head, All India Institute of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SKS/Med/Sleep_Preg
Record Dates: First submitted 2013-12-02; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Obstructive Sleep Apnea; Pregnancy Induced Hypertension; High-Risk Pregnancy; Restless Leg Syndrome; Infant, Very Low Birth Weight
Keywords: Obstructive Sleep Apnea in pregnancy; Pregnancy induced hypertension; Restless leg syndrome; Sleep
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension, Pregnancy-Induced; Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- polysomnography and AMBP on pregnant females (Experimental): Consecutive patients undergoing antenatal check up at the Antenatal Clinic at AIIMS hospital and obstetrics wards will be recruited and followed.Using Somnomedic systems, GmbH polysomnography machine by trained staff nurses and technicians at:
  Obstetrics ward, AIIMS hospital
  Interventions: Other: Polysomnography and ambulatory blood pressure recording

INTERVENTIONS:
Other: Polysomnography and ambulatory blood pressure recording

SUMMARY:
Hypothesis:Sleep Disorders are very common during pregnancy but the their exact role in causation of pregnancy related disorders is yet to be determined. OSA can complicate pregnancy given the risk factors of weight gain, upper displacement of the diaphragm, and hormonal-induced hyperaemia of the nasopharyngeal passages. SDB confers the risk of hypertensive disorders of pregnancy and is associated with adverse maternal and foetal outcomes.

The study would involve pregnant females which would be prospectively followed in pregnancy and post partum to know the prevalence of sleep disorders in pregnancy. Diagnosis of sleep disorders would be confirmed by overnight polysomnography and ambulatory blood pressure monitoring. Pregnancy outcomes, both maternal and fetal would be recorded and its relation with sleep disorders in pregnancy would be analysed.

DETAILED DESCRIPTION:
Objectives

1. To assess sleep quality during pregnancy
2. To know prevalence of various sleep disorders during pregnancy including restless leg syndrome, symptomatic obstructive sleep apnea etc.
3. To study the effect of sleep disorders on maternal and fetal outcome
4. To study the relation of obstructive sleep apnea with pregnancy induced hypertension.

Material & Methods

Study Design: Longitudinal prospective case-control study

* Consecutive patients undergoing antenatal check up at the Antenatal Clinic at AIIMS hospital during will be evaluated using questionnaires for sleep quality. Preliminary screening question for sleep disturbance in pregnancy to all patients
* Questionnaires used: Pittsburgh Sleep Quality Index (covers insomnia, RLS, snoring and sleep related breathing disorders); Epworth Sleepiness Score (for Excessive daytime sleepiness); Modified Wisconsin Score; Modified Berlin Questionnaires
* To now association between Obstructive sleep apnea and pregnancy induced hypertension patients who develop symptomatic OSA will be offered polysomnographic evaluation during the second/third trimester.
* An offer of similar services will be made to pregnant females who do not develop pregnancy induced hypertension at a similar gestational age.

Case: patient with OSA

Control: patients without OSA

* We proposed to determine that what proportion of the cases were exposed to sleep disorders and what proportion are not.
* We also planned to determine what proportion of controls is exposed and what proportion is not.

Cases and controls would be matched for age ,parity, BMI,previous h/o pre-eclampsia in first trimester.

Outcome parameters

1. Prevalence of various sleep disorders in pregnancy
2. Maternal outcome: Development of pregnancy induced hypertension (PIH), gestational diabetes mellitus, complicated pregnancy requiring admission, preterm delivery, ante-partum hemorrhage, delivery requiring intervention (Caesarian section, forceps/ventouse application)
3. Fetal outcome: APGAR scores at 1 and 5 min, IUGR, IUD, low birth weight

Sample Size:

A sample of convenience of 200 patients (who respond to questionnaire) and satisfy inclusion and exclusion criteria will be followed up prospectively to assess the effect of sleep disorders on pregnancy outcome.As per estimates from literature sample size for case control part would be 20 for cases and 40 controls.

Investigation specifically related to projects:

1. Using Somnomedic systems, GmbH polysomnography machine by trained staff nurses and technicians at:

   * Obstetrics ward, AIIMS hospital
   * Home based portable PSG in non admitted
2. Ambulatory blood pressure by the Oscar 2™ system from SunTech Medical, USA. The Oscar 2 is clinically validated to all three internationally recognized standards.

   * British Hypertension Society1 (A/A)
   * European Society of Hypertension International Protocol2
   * AAMI SP103

   Patient comfort The Oscar 2 and the Orbit™ BP cuff make patient comfort a priority.
   * The SunTech Medical, Inc. patented Orbit cuff uses an innovative stretch-sleeve design to maintain cuff placement and promote patient comfort.
   * The Oscar 2 is a light, compact monitor that uses motion tolerant algorithms to reduce re-inflates and failed readings. The auto-intelligent inflation pressure also reduces measurement time, promoting patient comfort by controlling cuff inflation.
3. Screening Polysomnography using Apnea linkTM PLUS

   * A quick and easy sleep-screening tool designed to help identify more patients at risk for obstructive sleep apnea (OSA).
   * A premium, compact device that can be used at home

Additional Investigation Required

* Routine clinical antenatal examination
* Blood pressure measurement
* Blood parameters (done routinely in ANC)

  * Fasting blood sugar
  * Renal and hepatic function tests
  * Hemoglobin levels/s ferritin
  * Serum TSH levels
* Urine examination

  * Routine and spot sample for protein.
* Sonography: To rule out twin pregnancy and molar gestation/IUGR/Anomalies.
* These investigations are routinely done in ante natal clinic at AIIMS.

Data Analysis

* Data will be collected on a pre-designed proforma.
* Statistical analysis will be performed using STATA 11 for Windows software (intercooled version, Stata Corporation, Houston, TX, USA).
* After assessing for approximate normal distribution, all continuous variables will be summarized as mean ± SD or median (interquartile range).
* Categorical variables will be expressed as n (%).
* The cases and controls will be compared using unpaired t-test if the data was normally distributed and the Mann-Whitney U test if not.
* A p values of <0.05 will be considered statistically significant.
* Confounding factors influencing pregnancy outcomes will be subject to multivariate analysis to determine significance.

ELIGIBILITY:
Inclusion criteria

* Age 20-45 years
* Singleton pregnancy

Exclusion criteria

* Known hypertensives i.e SBP>140/DBP>90/on anti-hypertensive medications prior to pregnancy
* Known diabetics (FBS>100, 75 g OGTT positive/on medications)
* Hypothyroidism
* Chronic renal failure
* Chronic liver disease
* Twin pregnancy
* Known systemic inflammatory condition e.g APLA Syndrome,SLE
* Molar gestation
* Patients on nephrotoxic medications e.g.NSAIDS
* Exclusion criteria for case control part only.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Sleep quality in pregnancy and its association with pregnancy outcomes | from recruitment during pregnancy to 6 weeks post partum

SECONDARY OUTCOMES:
Number of patients who develop PIH and gestational diabetes | from recruitment to 6 weeks post partum

OTHER OUTCOMES:
to know the prevalence of sleep disorders in pregnancy and post partum | from recruitment in pregnancy to 6 week post partum

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K Sharma, MD, Ph.D., Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, New Delhi, India